CLINICAL TRIAL: NCT05063890
Title: Comparison of Muscle Specific and Movement Specific Muscle Energy Technique in the Management of Mechanical Neck Pain: a Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2021/6
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Neck Pain
Keywords: neck pain
MeSH Terms: conditions — Neck Pain | interventions — Heating; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Specific MET (Experimental)
  Interventions: Procedure: Muscle Specific Post Isometric Relaxation MET; Procedure: unilateral postero-anterior glide; Procedure: Heating and TENS
- Movement specific MET (Experimental)
  Interventions: Procedure: Movement Specific Post Isometric Relaxation MET; Procedure: unilateral postero-anterior glide; Procedure: Heating and TENS

INTERVENTIONS:
Procedure: Muscle Specific Post Isometric Relaxation MET — 3-5 reps of Post Isometric Relaxation MET targeted at muscles of the neck prone to get short
  Arms: Muscle Specific MET
Procedure: Movement Specific Post Isometric Relaxation MET — 3-5 reps of Post Isometric Relaxation MET targeted at specific movements of the cervical spine
  Arms: Movement specific MET
Procedure: unilateral postero-anterior glide — 3 sets of unilateral posteroanterior glide (10-15 oscillations) at the involved segment
Procedure: Heating and TENS — Heating and TENS for 10 minutes

SUMMARY:
the purpose of this study is to compare the effects of muscle-specific muscle energy technique and movement-specific muscle energy technique in terms of pain, function and cervical range of motion in persons with mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

Mechanical neck pain ranging from 40-80 mm on visual analogue scale (VAS) Age between 19-44 years Pain or limitation on cervical motion

-

Exclusion Criteria:

History of fracture, surgery or trauma in the neck Cervical radiculopathy Myelopathy Spondylosis Syringomyelia Thoracic outlet syndrome Infection Malignancy Inflammatory or rheumatic disorders Vascular syndromes

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 5 days
  Pain will be measured using Visual Analogue Scale, with greater score signifying greater pain
Neck Disability Index | 5 days
  Function and neck related disability will be measured using Neck Disability Index, with greater score signifying greater disability and poorer outcome
Cervical Range of Motion | 5 days
  Cervical Range of Motion will be measured using a universal goniometer, with greater score signifying more favorable outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No